CLINICAL TRIAL: NCT00079885
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Comparative Study Of The Efficacy And Safety Of Tigecycline Vs Levofloxacin To Treat Subjects Hospitalized With Community-Acquired Pneumonia
Brief Title: Study Evaluating Tigecycline vs Levofloxacin in Hospitalized With Community-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 3074A1-308
Record Dates: First submitted 2004-03-18; First posted 2004-03-19 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Community Acquired Pneumonia; Bacterial Pneumonia; Cross Infection
Keywords: Bacterial Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia, Bacterial; Cross Infection | interventions — Tigecycline

INTERVENTIONS:
Drug: tigecycline

SUMMARY:
To compare the efficacy and safety of tigecycline with those of levofloxacin in the treatment of subjects with CAP requiring hospitalization. The co-primary efficacy endpoints in the study will be the clinical response in the clinically evaluable population and the clinical response in the clinical modified intent-to-treat population at the TOC visit. The primary efficacy analyses will first determine whether tigecycline is noninferior to levofloxacin. If tigecycline is found to be noninferior, the analyses will determine whether tigecycline is statistically better than levofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years of ag.
* Subjects hospitalized with CAP for whom IV antibiotic treatment is indicated
* The presence of fever (within 24 hours prior to randomization), defined as oral temperature >38°C/100.4°F, axillary temperature >38.1°C/100.6°F, tympanic temperature >38.5°C/ 101.2°F, or a rectal/core temperature >39°C/102.2°F OR hypothermia (within 24 hours prior to randomization), core temperature <35°C/95°

Exclusion Criteria:

* Any concomitant condition that, in the opinion of the investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy could be completed (eg, life expectancy <30 days)
* Hospitalization within 14 days prior to the onset of symptoms
* Residence in a long-term care facility or nursing home ≥14 days before the onset of symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2003-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Bergallo C, Jasovich A, Teglia O, Oliva ME, Lentnek A, de Wouters L, Zlocowski JC, Dukart G, Cooper A, Mallick R; 308 Study Group. Safety and efficacy of intravenous tigecycline in treatment of community-acquired pneumonia: results from a double-blind randomized phase 3 comparison study with levofloxacin. Diagn Microbiol Infect Dis. 2009 Jan;63(1):52-61. doi: 10.1016/j.diagmicrobio.2008.09.001. Epub 2008 Nov 5. PMID 18990531
- [Derived] Tanaseanu C, Bergallo C, Teglia O, Jasovich A, Oliva ME, Dukart G, Dartois N, Cooper CA, Gandjini H, Mallick R; 308 Study Group; 313 Study Group. Integrated results of 2 phase 3 studies comparing tigecycline and levofloxacin in community-acquired pneumonia. Diagn Microbiol Infect Dis. 2008 Jul;61(3):329-38. doi: 10.1016/j.diagmicrobio.2008.04.009. Epub 2008 May 27. PMID 18508226